CLINICAL TRIAL: NCT01382524
Title: Peripheral I.V. Catheter Complication Rate Comparison of Two Different Catheter-Stabilization Systems
Brief Title: Peripheral Intravenous Catheter Complication Rate Comparison of Two Different Catheter-Stabilization Systems
Acronym: PIV Secural
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-011427
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Catheter Complications
Keywords: PIV therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stabilization system A: A commercialized stabilization dressing using a winged PIV catheter.
- Stabilization System B: A commercialized stabilization device using a non-winged PIV catheter

SUMMARY:
Approximately 300 million short peripheral intravascular catheters (PIVs) were sold in the U.S. in 2009. These short (< 3 inches) peripherally inserted IV catheters are vital for providing patients with needed: 1) fluid, electrolyte, nutrient and blood product replacement, 2) medicines and 3) diagnostic solutions (dyes). However, these IV catheters have inherent risks or potential complications which may result from poor catheter securement or stabilization.

When a PIV catheter is not properly secured, motion and micro-motion within the vessel cause injury to the vein. This damage to the vein is a primary cause of phlebitis, a distressing complication of PIV therapy. Additional complications of inadequate stabilization of the PIV catheter are infiltration, leaking at the insertion site, pain, infection and dislodgement. According to Royer (2003), the most common reason for PIV catheter failure is infiltration and dislodgement. Infiltration is more dependent on keeping the extremity still, where phlebitis is dependent on injuries due to the chemical nature of the drugs and fluids infused or by the physical trauma to the endothelium from IV pushes.

The results of these complications are costly and can be serious if another vein cannot be immediately accessed or if the infiltrated infusate causes tissue necrosis. An unscheduled restart of another PIV catheter causes a delay in patient treatment, patient discomfort, patient dissatisfaction, safety concerns, nursing interruptions and additional costs. Actual costs associated with PIV catheter restarts include materials and nursing resources; yet intangibles such as, treatment for patient complications and patient dissatisfaction may be far more costly.

One way to reduce the incidence of PIV catheter-associated complications is to use technologies that help reduce catheter movement thereby improving catheter stabilization. In addition to stabilization platforms added to the peripheral IV catheter design, catheter stabilization devices and modified transparent film dressings also help to reduce catheter movement and could possibly eliminate the need for routine catheter site changes.

Therefore, the purpose of this study is to: 1) compare the number of PIV securement-related complications and PIV catheter restarts of one stabilization system to another stabilization system and 2) to determine which system provides a cost savings.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, unless an emancipated minor
* A patient who is admitted or going to be admitted to the hospital
* Requires peripheral IV therapy (catheter) for an anticipated 72 hours or longer.
* Has an insertion site in the forearm or hand free of deformities, phlebitis, infiltration, dermatitis, burns, lesions or tattoos
* Demonstrates cooperation with a catheter insertion and the securement protocol.

Exclusion Criteria:

* Is a current participant or a past participant in this study
* If the study PIV catheter will cross a joint or the catheter hub will hang off the fingers
* If the study PIV catheter site will be placed below an old infusion site
* If the study PIV site needs to be immobilized with a splint or other devices
* Has a documented or a known allergy or sensitivity to a medical adhesive product such as transparent film adhesive dressings, tapes or liquid skin protectants
* Requires the application of a gauze pad, a topical ointment or solution under the dressing in addition to the prep(s) required in the protocol
* Has or has had a previous IV catheter related phlebitis or infiltration during this hospitalization.
* Will have a vesicant administered through the study catheter, e.g. Dilantin
* Will require a power injection for a radiologic procedure during participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study will be male and female patients who are at least 18 years of age or an emancipated minor, require a peripheral IV catheter for an anticipated three days (72 hours) or longer
Sampling Method: Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
PIV Catheter complication rates | Anticipated to be up to 4 days per participant
  The primary endpoint for the study is the difference between the number and type of PIV-related complications (phlebitis, infiltration, dislodgement, leakage, local site infection and catheter line associated infection) between the two stabilization groups.

SECONDARY OUTCOMES:
Cost effectiveness | Anticipated to be up to 4 days per participant
  The secondary endpoints are overall and specific complication rates, incidence of unscheduled restarts, incremental cost effective ratio for one stabilization system to another stabilization system.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Coombs, MD, Principal Investigator — University of North Carolina, Chapel Hill; Cedric Lefebvre, MD, Principal Investigator — Wake Forest University
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina